CLINICAL TRIAL: NCT04862520
Title: Prognostic Factors for Work Disability in Patients With Chronic Widespread Pain and Fibromyalgia: Protocol for a Cohort Study
Brief Title: Prognostic Factors for Work Disability in Patients With Chronic Widespread Pain and Fibromyalgia.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Henning Bliddal, Professor, Frederiksberg University Hospital
Other Study IDs: PDH4
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Chronic Widespread Pain; Fibromyalgia
MeSH Terms: conditions — Chronic Pain; Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction:

The association between chronic widespread pain (CWP) and disability is well-established. Although research support large inter-individual differences in functional outcomes, limited studies are available on the socio-economic consequences of offering stratified treatment based on prognostic factors. Identification of predictors of long-term functional outcomes such as work disability as a critical consequence, could assist early and targeted personalised interventions. The primary objective of this cohort study is to identify prognostic factors for the primary endpoint work status (employed and working vs not working) in patients with CWP assessed 3- years from baseline, i.e. at referral for specialist care.

Methods and analyses:

Data are collected at the diagnostic unit at Department of Rheumatology, Frederiksberg Hospital. The first 1,000 patients >=18 years of age registered in a clinical research database (DANFIB registry) with CWP either "employed and working" or "not working" will be enrolled. Participants must meet the American College of Rheumatology (ACR) 1990 definition of CWP, i.e. pain in all four body quadrants and axially for more than three months and are additionally screened for fulfilment of criteria for FM. Clinical data and patient-reported outcomes are collected at referral (baseline) through clinical assessment and electronic questionnaires. Data on the primary endpoint work status at baseline and 3- years from baseline will be extracted from the Integrated Labour Market Database, Statistics Denmark and the nationwide Danish DREAM database. Prognostic factor analysis will be based on multivariable logistic regression modelling with the dichotomous work status as dependent variable.

DETAILED DESCRIPTION:
By using prognostic factor research, the purpose is to understand and improve future outcomes in patients with CWP. Identification of prognostic factors for long-term functional outcomes, including work disability, could assist tailoring and timing the therapeutic decision for specific patients and potentially optimise functional outcomes compared with offering standardised (i.e. ignorant) intervention programs to patients with CWP.

The results from this cohort study are anticipated to contribute with relevant knowledge that may be used to guide future intervention matching and delivery of stratified interventions based on prognostic classification.

Study design:

The study is designed as a clinical cohort study enabling multivariable logistic regression modelling of data from the large Danish DANFIB cohort of CWP patients with the primary aim assessed after 3- years.

Setting:

Data collection takes place in a specialised clinical care setting at the diagnostic unit at Department of Rheumatology, Frederiksberg Hospital. Here patients presenting with CWP, either as their primary pain problem or secondary to other established rheumatic disease, have been offered clinical assessment and screening for CWP since 1st of January 2018.

The electronic data collection is accessed via touchscreens and data are exported to a designated clinical research database (the DANFIB registry). Data extracted from electronic patient files, including findings at clinical examination (manual TP count), are also integrated into the DANFIB registry. A protocol outlining the content and objectives of the DANFIB registry can be accessed online.The DANFIB registry will serve as point of departure for the current cohort study.

Participants:

The first 1,000 patients consecutively registered in the DANFIB registry with CWP independent of working status. Participant inclusion is expected to be completed by December 2021. Informed consent will be obtained for all participants when registered in the DANFIB registry.

Data sources:

Baseline demographics, clinical characteristics and individual labour market status assessed at baseline will be extracted from the DANFIB registry. Data on the primary endpoint work status ("employed and working" or "not working") at baseline and again 3- years from baseline will be extracted from the Integrated Laboure Market Database at Statistics Denmark and the nationwide Danish DREAM database.

ELIGIBILITY:
Inclusion Criteria:

participants must:

* be over 18 years of age
* able to understand and read Danish
* have retrievable data in the DANFIB registry

Exclusion Criteria:

* no consent
* do not read and understand Danish
* non-retrievable data in the DANFIB registry
* any form of pension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic widespread pain (CWP) is prevalent in the background population with an estimated prevalence of about 10% and represents a major clinical challenge due to the complexity of the disease. Apart from pain and other centrally mediated symptoms, CWP is strongly associated with disability affecting activities of daily living (ADL), incapacity for normal employment and poor social participation. Fibromyalgia (FM) is the best characterised subset of patients presenting with CWP and is by many considered to represent the upper end of a pain severity spectrum, i.e. associated with greater disease burden and higher levels of disability, in comparison to patients with CWP not fulfilling FM disease criteria or more localized pain conditions.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Work status on the overall cohort | 3 years
  To reveal prognostic factors, among the cohort of CWP patients, that are associated with the primary endpoint work status (employed and working vs not working) assessed after 3- years.

SECONDARY OUTCOMES:
Work status on those employed and working at baseline | 3 years
  Identification of prognostic factors for work status (employed and working vs not working) after 3- years in patients with CWP, who are employed and working at baseline.
Work status on those not working at baseline | 3 years
  III. identification of prognostic factors for work status (employed and working vs not working) after 3- years in patients with CWP, who are not working at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Pernille H. Duhn, dr., Study Chair — Parker Institute
Locations (1):
- Frederiksberg Hospital, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duhn PH, Locht H, Waehrens EE, Christensen R, Thielen K, Henriksen M, Kristensen LE, Bliddal H, Amris K. Prognostic factors for work disability in patients with chronic widespread pain and fibromyalgia: protocol for a cohort study. BMJ Open. 2021 Dec 22;11(12):e052919. doi: 10.1136/bmjopen-2021-052919. PMID 34937720